CLINICAL TRIAL: NCT02232139
Title: Measurement of Psychomotor Function Recovery in Patients After General Anesthesia Using 4-Choice Reaction Time Test
Brief Title: Measurement of Psychomotor Recovery After Anesthesia Using 4CRT
Acronym: 4CRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Department of Anesthesiology, Hospital Dresden-Friedrichstadt, Dresden, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BR-87/13-1; EK-BR-87/13-1 (Other: Ethics commission)
Record Dates: First submitted 2014-08-28; First posted 2014-09-05 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Delayed Recovery From Anaesthesia
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard therapy group (No Intervention): Participant who will not receive midazolam for pharmacological anxiolytic premedication before general surgery
- Midazolam group (Experimental): Participant who will receive midazolam for pharmacological anxiolytic premedication before general surgery
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — The participants receive the pharmacological premedication before the surgery anyway
  Other Names: Dormicum
  Arms: Midazolam group

SUMMARY:
The aim of the investigation is to validate the SmartPhone-based 4-Reaction Choice Time Test (4CRT) as a measure for recovery of the psychomotor function in patients after general anesthesia. One hundred female patients, scheduled to ambulatory gynecological surgery in general anesthesia, will be randomized to the group with pharmacological anxiolytic premedication with midazolam (N=50) and to the group without midazolam (N=50). All patients will be monitored using 4CRT before and after standardized general anesthesia. The reaction time, measured with 4CRT is the primary outcome parameter of the investigation.

DETAILED DESCRIPTION:
4CRT is a classical psychological test, used to measure the psychomotor speed. This test measures choice reaction time. The participants are instructed to respond by pressing the keys 1-4 of the keyboard, corresponding to the numbers, appearing on the screen of computer (PDA, SmartPhone). The average of the response latency, measured during the 10 trials is usually taken as 4CRT outcome.

ELIGIBILITY:
Inclusion Criteria:

* Physical status I-III according to American Society of Anesthesiology
* ambulatory gynecologic surgery of 10-40 min
* patient is able to use VAS and to use SmartPhone-based 4CRT
* given informed consent

Exclusion Criteria:

* age < 18 or > 50 years
* patients who are not able to give their informed consent
* surgery lasts more than 40 min.
* history of psychopharmaceuticals or analgesics

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Change of four choice reaction time from baseline | One time before the surgery and 2 hours after the surgery
  One time immediately before the surgery and 6 times within 2 hours after the surgery for each participant

SECONDARY OUTCOMES:
Concentration of midazolam in serum | Within 2 hours after the surgery only in 40 (20 from each group) participants

OTHER OUTCOMES:
Postanesthesia discharge scoring system | Within 2 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Taras I Usichenko, MD, PhD, Study Director — University Medicine of Greifswald
Locations (1):
- Department of Anesthesiology, Intensive Care Medicine, Emergency Medicine and Pain Therapy, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zuurmond WW, Balk VA, van Dis H, van Leeuwen L, Paul EA. Multidimensionality of psychological recovery from anaesthesia. Analysing six recovery tests. Anaesthesia. 1989 Nov;44(11):889-92. doi: 10.1111/j.1365-2044.1989.tb09141.x. PMID 2596654